CLINICAL TRIAL: NCT05121987
Title: Analgesic and Respiratory Outcomes in Patients Receiving Continuous Bilateral Erector Spinae Plane Block Compared to Continuous Preperitoneal Catheter Wound Infusion After Upper Abdominal Surgery: a Randomized Double-blind Study
Brief Title: Analgesic and Respiratory Outcomes in Patients Receiving Continuous Bilateral Erector Spinae Plane Block Compared to Continuous Preperitoneal Catheter Wound Infusion After Upper Abdominal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: South Egypt Cancer Institute (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abd El-Hameed Osman, Assistant lecturer, South Egypt Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 563
Record Dates: First submitted 2021-11-04; First posted 2021-11-16 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Abdominal Cancer Surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Erector spinae plane block (Active Comparator)
  Interventions: Procedure: Erector Spinae Plane block
- Continuous wound infusion (Active Comparator)
  Interventions: Procedure: Continuous Wound Infusion

INTERVENTIONS:
Procedure: Erector Spinae Plane block — An ultrasound linear probe is going to be placed in a longitudinal orientation 3 cm lateral to the T6 spinous process corresponding to the T5 transverse process. . Local infiltration with 2% of lignocaine at the site of needle insertion is going to be administered. Using in plane approach an 18 G Tuohy needle will be inserted in caudal-cephalad direction, until the tip is deep to erector spinae muscle, as evidenced by visible hydro-dissection below the muscle plane, and on injection of 5 ml of normal saline.
  Arms: Erector spinae plane block
Procedure: Continuous Wound Infusion — Towards the end of surgery, a multiholed 15-cm Anesthesia catheter will be placed in the preperitoneal space (the subfascial space between the peritoneum and posterior fascia) under direct vision and to be tunneled via the rectus sheath to the skin, rolled out and exiting laterally and stabilized with an adhesive tape on skin.
  Arms: Continuous wound infusion

SUMMARY:
We aim to compare the postoperative analgesic and respiratory outcomes in patients receiving continuous bupivacaine infusion via bilateral erector spinae catheters versus preperitoneal catheters in upper abdominal surgeries.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II, weighing 50-90 Kg with Body Mass Index (BMI) 18.5- 29.9 kg/m2

Exclusion Criteria:

* ASA physical status ≥III, pregnancy, body mass index >30 kg/m2, preoperative opioid consumption, patient's refusal and contraindications of the use of spirometry or either of the truncal blocks under the study including; respiratory, cardiac, neurological, mental or coagulation disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Total Morphine consumption | 48 hours

IPD SHARING:
Plan to Share IPD: Undecided